CLINICAL TRIAL: NCT02054637
Title: Resolving Bile Reflux by Lanreotide in Patients With Roux-en-Y Gastrojejunostomy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Kim Moubax, Dr. Kim Moubax, gastro-enterology, Universitair Ziekenhuis Brussel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PHV106-B.05
Record Dates: First submitted 2014-01-29; First posted 2014-02-04 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-01

CONDITIONS: Acid Reflux Esophagitis; Non-acid Reflux Esophagitis
Keywords: Bile reflux; Reflux esophagitis; Lanreotide autogel; Somatuline; Endoscopy; Impedancemetry
MeSH Terms: conditions — Bile Reflux; Esophagitis, Peptic | interventions — lanreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lanreotide (Experimental): Lanreotide autogel 120mg injection every 4 weeks (every patient will receive 3 injections)
  Interventions: Drug: Lanreotide

INTERVENTIONS:
Drug: Lanreotide
  Other Names: Somatuline

SUMMARY:
Somatostatine induces a dose-dependent reduction of postprandial plasma cholecystokinin (CCK) secretion with a concomitant inhibition of postprandial gallbladder contraction, abolishing almost completely bile salts output from the gallbladder. Somatostatine is also known to decrease acid production with significant increase of intragastric pH. In this way, somatostatine could influence acid as well as non-acid reflux by decreasing gallbladder emptying and decreasing acid secretion.

Purpose of the study is to evaluate the efficacy of lanreotide autogel 120 mg on symptoms and endoscopic lesions in patients with an endoscopic gastrointestinal reflux esophagitis that cannot be controlled with classic therapy.

DETAILED DESCRIPTION:
Patients presenting with persistent esophagitis on endoscopy while on proton pump inhibitors (PPI) treatment will receive a maximal therapy consisting of 2 x 40 mg of PPI before the meals (morning and evening) and a H2 blocker before bedtime (standard practice). They will be reevaluated endoscopically and clinically 2 months later (standard practice). If reflux persists, objectivized by impedancemetry (standard practice), they will be asked to participate in this study.

Lanreotide autogel 120 mg deep subcutaneously every 4 weeks will be added to the treatment. A total of 3 injections per patient have been foreseen in this proof of concept study.

Patients will be reevaluated clinically after 2, 4 and 8 weeks. At the end of the study a new upper gastrointestinal endoscopy and impedancemetry will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Persistent endoscopic reflux in spite of maximal medical therapy with PPI 2 x 40 mg (before breakfast and dinner) and 300 mg of H2 blocker ranitidine (at bedtime).

The Los Angeles classification (LA) will be used to evaluate endoscopic reflux. Any distal esophageal ulcer with negative biopsy is also diagnostic for reflux.

Persistent reflux is defined as:

No reflux complaints but continuing endoscopic lesions and positive impedancemetry.

Reflux complaints with continuing endoscopic lesions and positive impedancemetry.

Reflux complaints without endoscopic lesions but positive impedancemetry.

Exclusion Criteria:

* Pregnancy or inadequate anticonception, breast feeding.
* Negative impedancemetry.
* Diabetes.
* Placement of a gastric ring for weight loss.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-12 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Los Angeles criteria for reflux esophagitis | 4 weeks after the last injection with lanreotide
  Endoscopy at the start of the study will be compared with endoscopy at the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Kim Moubax, Assistent, Study Chair — University hospital of Brussels, Laarbeeklaan, Jette
Locations (1):
- University Hospital of Brussels, Jette, Belgium

REFERENCES:
- [Background] Ishikawa M, Kitayama J, Kaizaki S, Nakayama H, Ishigami H, Fujii S, Suzuki H, Inoue T, Sako A, Asakage M, Yamashita H, Hatono K, Nagawa H. Prospective randomized trial comparing Billroth I and Roux-en-Y procedures after distal gastrectomy for gastric carcinoma. World J Surg. 2005 Nov;29(11):1415-20; discussion 1421. doi: 10.1007/s00268-005-7830-0. PMID 16240061
- [Background] Montesani C, D'Amato A, Santella S, Pronio A, Giovannini C, Cristaldi M, Ribotta G. Billroth I versus Billroth II versus Roux-en-Y after subtotal gastrectomy. Prospective [correction of prespective] randomized study. Hepatogastroenterology. 2002 Sep-Oct;49(47):1469-73. PMID 12239969
- [Background] Gerard PS, Gerczuk P, Finestone H. Bile reflux in the esophagus demonstrated by HIDA scintigraphy. Clin Nucl Med. 2007 Mar;32(3):224-5. doi: 10.1097/01.rlu.0000255039.24698.48. No abstract available. PMID 17314604
- [Background] Swartz DE, Mobley E, Felix EL. Bile reflux after Roux-en-Y gastric bypass: an unrecognized cause of postoperative pain. Surg Obes Relat Dis. 2009 Jan-Feb;5(1):27-30. doi: 10.1016/j.soard.2008.10.009. Epub 2008 Oct 30. PMID 19095503
- [Background] Gans SL, van Westreenen HL, Kiewiet JJ, Rauws EA, Gouma DJ, Boermeester MA. Systematic review and meta-analysis of somatostatin analogues for the treatment of pancreatic fistula. Br J Surg. 2012 Jun;99(6):754-60. doi: 10.1002/bjs.8709. Epub 2012 Mar 20. PMID 22430616
- [Background] Drewe J, Sieber CC, Mottet C, Wullschleger C, Larsen F, Beglinger C. Dose-dependent gastrointestinal effects of the somatostatin analog lanreotide in healthy volunteers. Clin Pharmacol Ther. 1999 Apr;65(4):413-9. doi: 10.1016/S0009-9236(99)70136-0. PMID 10223779
- [Background] Lamrani A, Vidon N, Sogni P, Nepveux P, Catus F, Blumberg J, Chaussade S. Effects of lanreotide, a somatostatin analogue, on postprandial gastric functions and biliopancreatic secretions in humans. Br J Clin Pharmacol. 1997 Jan;43(1):65-70. doi: 10.1111/j.1365-2125.1997.tb00034.x. PMID 9056054
- [Background] Ludlam WH, Anthony L. Safety review: dose optimization of somatostatin analogs in patients with acromegaly and neuroendocrine tumors. Adv Ther. 2011 Oct;28(10):825-41. doi: 10.1007/s12325-011-0062-9. Epub 2011 Sep 28. PMID 21964965